CLINICAL TRIAL: NCT01317446
Title: Effect of an Amine Fluoride/Stannous Fluoride Containing Mouthrinse on Gingival Inflammation,Plaque Development, Discoloration and Bacterial Plaque Composition Over Six Months.
Brief Title: Effect of Mouthrinsing on Inflammation of the Gums.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Gaba International AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GASAS-1007X
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Gingivitis
Keywords: gingivitis index; plaque index; discoloration index; mouth rinse; amine fluoride/stannous fluoride; clinical trial
MeSH Terms: conditions — Gingivitis | interventions — Tin Fluorides; Meridol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- amine fluoride/stannous fluoride (Experimental): Amine fluoride/stannous fluoride mouthrinse in addition to mechanical oral hygiene
  Interventions: Drug: amine fluoride/stannous fluoride
- No rinsing (No Intervention): Mechanical oral hygiene only

INTERVENTIONS:
Drug: amine fluoride/stannous fluoride — 10 ml qd, oral, topical, 6 months duration
  Other Names: meridol
  Arms: amine fluoride/stannous fluoride

SUMMARY:
The purpose of this study is to determine whether rinsing with an amine fluoride/stannous flouride mouthrinse in addition to daily tooth brushing is more effective than tooth brushing alone.

DETAILED DESCRIPTION:
Gingivitis prevalence is 100% among the population. This is mostly due to an inadequate mechanical cleaning of the teeth. However, remaining dental biofilm can be approached by antibacterial mouthrinses. As a consequence of regular use of these mouthrinses, gingivitis can be reduced. Amine fluoride/stannous flouride mouthrinse (ASF)has proved its efficacy in several studies. In the previous years, a new formulation that does not contain ethanol anymore was introduced in the market. Therefore, it is the aim of the study to proof whether rinsing with ASF adjunctive to mechanical oral hygiene is more effective on gingivitis reduction than mechanical oral hygiene alone. In addition, effects on dental plaque, discoloration of teeth and bacterial colonization should be studied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults aged ≥18 years.
* Participants who have gingivitis/mild chronic periodontitis (approximal probing depth ≤ 3.5 mm at ≥ 80 % of the sites and at ≤ 20 % of the sites > 3.5 mm and < 5 mm).
* Participants must have read, understood and signed the informed consent form.
* Participants who have a GI ≥ 1.3 at baseline.
* Participants who have at least 20 own teeth excluding the wisdom teeth (incl. 16 natural crowns).
* Participants who have an acceptable compliance according to the investigators' assessment.

Exclusion Criteria:

* Participants who have systemic diseases that require regular systemic medication intake that may affect the gingival condition (e. g. phenytoin, nifedipine, cyclosporine, antibiotics, steroids, antiphlogistics).
* Participants who require antibiotic treatments for dental appointments (endocarditis prophylaxis).
* Participants who were treated with antibiotics 8 weeks before recruitment and during the course of the study.
* Participants who were treated with any antibacterial mouthrinse 6 weeks before recruitment.
* Participants who use other than the recommended mouthrinse or toothpaste during the study period.
* Participants who have moderate and severe chronic or aggressive periodontitis.
* Participants who have irregularities of the gingival tissues, e. g. hyperplastic gingiva, mucosal diseases.
* Participants who have rampant caries.
* Participants under guardianship or without freedom by administrative or legal award.
* Known hypersensitivity or allergy to the study product and standard toothpaste ingredients used in the present study.
* Known pregnancy or breast feeding during the course of the study.
* Participation in another clinical trial or receipt of an investigational compound/treatment at the same time and 4 weeks prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Reduction in gingivitis | 6 months
  To proof whether rinsing with ASF adjunctive to mechanical oral hygiene is more effective on gingivitis reduction than mechanical oral hygiene alone.

SECONDARY OUTCOMES:
Reduction in plaque | 6 months
  To proof whether rinsing with ASF adjunctive to mechanical oral hygiene is more effective on plaque reduction than mechanical oral hygiene alone.
Discoloration of teeth | 6 months
  To proof the effect of rinsing with ASF on discoloration of teeth
Bacterial colonization | 6 months
  To proof whether rinsing with ASF adjunctive to mechanical oral hygiene influences bacterial colonization
Adverse events | 6 months
  Recording all adverse events over the entire rinsing period

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hoffmann, Prof. Dr., Principal Investigator — Technische Universität Dresden
Locations (1):
- Dreden University of Technology, Universitätsklinikum, Poliklinik für Parodontologie, Dresden, Saxony, Germany